CLINICAL TRIAL: NCT02197975
Title: A Phase I, Randomized, Double Blind, Placebo-Controlled, Two Period, Ascending Dose, Crossover Study to Assess the Safety and Pharmacokinetics of Two Doses of PT010 in Healthy Adult Subjects of Japanese Descent Following a Single Dose and After Chronic Dosing for 7 Days
Brief Title: Randomized, Crossover Safety and Pharmacokinetics Study of PT010
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT010003-00
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: COPD
Keywords: Healthy Volunteers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PT010 Dose 1 (Experimental): PT010 Dose 1; Budesonide, Glycopyrrolate, and Formoterol Fumarate (BGF) Inhalation Aerosol. Administered as 2 inhalations.
  Interventions: Drug: PT010 Dose 1
- PT010 Dose 2 (Experimental): PT010 Dose 2; Budesonide, Glycopyrrolate, and Formoterol Fumarate (BGF) Inhalation Aerosol. Administered as 2 inhalations.
  Interventions: Drug: PT010 Dose 2
- Placebo MDI (Placebo Comparator): Placebo MDI. Administered as 2 inhalations
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: PT010 Dose 1 — PT010 Dose 1; Budesonide, Glycopyrrolate, and Formoterol Fumarate (BGF) Inhalation Aerosol. Administered as 2 inhalations.
  Arms: PT010 Dose 1
Drug: PT010 Dose 2 — PT010 Dose 2; Budesonide, Glycopyrrolate, and Formoterol Fumarate (BGF) Inhalation Aerosol. Administered as 2 inhalations.
  Arms: PT010 Dose 2
Drug: Placebo MDI — Placebo MDI. Administered as 2 inhalations
  Arms: Placebo MDI

SUMMARY:
Safety and Pharmacokinetics of Two Doses of PT010 in Healthy Adult Subjects of Japanese Descent Following a Single Dose and After Chronic Dosing for 7 Days.

DETAILED DESCRIPTION:
This is a Phase I, single-center, randomized, double-blind, placebo-controlled, two period, ascending dose, cross-over study to assess safety and PK of two doses of PT010 in healthy adult subjects of Japanese descent. Safety and PK will be assessed following a single dose and during twice-daily (BID) chronic dosing for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent Form (ICF) prior to any study related procedures
* Male and female subjects first generation Japanese subjects 18 to 55 years, inclusive
* Body weight ≥50 kg (110 lbs) at the Screening Visit and body mass index between 18.5 and 32 kg/m2, inclusive
* Good general health
* Medically acceptable contraception for women of child-bearing potential and males with female partners of childbearing potential
* Clinical labs within normal ranges or determined to be not clinically significant by the Investigator

Exclusion Criteria:

* Pregnancy, nursing female subjects, or subjects trying to conceive
* Clinically significant neurologic, cardiovascular, hepatic, renal, endocrinologic, pulmonary, hematological, psychiatric, or other medical illness that would interfere with participation in this study
* History of ECG abnormalities
* Cancer not in complete remission for at least 5 years
* Clinically significant, symptomatic prostatic hypertrophy
* Male subjects with a trans-urethral resection of the prostate or full resection of the prostate within 6 months prior to Screening
* Clinically significant bladder neck obstruction or urinary retention
* Inadequately treated glaucoma
* History of an allergic reaction or hypersensitivity to any drug or to any component of the formulations used in this study
* Subjects with pre-existing anemia and/or iron deficiency

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic profile of PT010 | 12 hours
  The pharmacokinetic profile of PT010 will be assessed at the first day (Day 1) and last dose (Day 8) in each Treatment Period based on:
  * maximum plasma concentration (Cmax)
  * area under the plasma concentration-time curve from 0 to 12 hours (AUC0 12)
  * area under the plasma concentration-time curve from 0 to the time of the last measureable plasma concentration (AUC0-t)
  * area under the plasma concentration-time curve from 0 extrapolated to infinity (AUC0-∞) (only calculated for Day 1)
  * time to maximum plasma concentration (tmax)
  * apparent terminal elimination half-life (t½)
  * apparent total body clearance (CL/F)
  * apparent volume of distribution (Vd/F)
  * terminal elimination rate constant (λz)
  * accumulation ratio for Cmax (RAC [Cmax])
  * accumulation ratio for AUC0 12 (RAC [AUC0 12]) Other PK parameters may be calculated, as appropriate.

SECONDARY OUTCOMES:
Overall safety of PT010 | 12 hours
  The safety associated with the use of PT010 will be assessed from physical examination findings, adverse event (AE) reporting, vital signs, clinical laboratory values, and findings from 12 lead electrocardiograms (ECGs).

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Orevillo, Study Chair — Pearl Therapeutics
Locations (1):
- SNBL Clinical Pharmacology Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Huang Y, Assam PN, Feng C, Su R, Dorinsky P, Gillen M. Ethnic pharmacokinetic comparison of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler (BGF MDI) between Asian and Western healthy subjects. Pulm Pharmacol Ther. 2020 Oct;64:101976. doi: 10.1016/j.pupt.2020.101976. Epub 2020 Nov 2. PMID 33152467